CLINICAL TRIAL: NCT01770977
Title: Effects of Phototherapy by Light-emitting Diode Therapy (LEDT) on Clinical, Biochemical and Biomechanical of Muscle Performance in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Centro de Pequisas de Ótica e Fotônica (Other)
Responsible Party: Principal Investigator, Cleber Ferraresi, MSc, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE: 0327.0.135.000-11
Record Dates: First submitted 2012-09-15; First posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2012-09

CONDITIONS: Athlete
Keywords: Light-emitting diode therapy; Muscle performance; Aerobic performance; Lactate; Creatine kinase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Effective Light-emitting diode therapy (Active Comparator): Effects of light-emitting diode therapy on clinical, biochemical and biomechanical of muscle performance in athletes
  Interventions: Device: Light-emitting diode therapy
- Placebo light-emitting diode therapy (Placebo Comparator): Effect of placebo light-emitting diode therapy on clinical, biochemical and biomechanical of muscle performance in athletes
  Interventions: Device: Placebo light-emitting diode therapy

INTERVENTIONS:
Device: Light-emitting diode therapy
  Other Names: LED; LED therapy
  Arms: Effective Light-emitting diode therapy
Device: Placebo light-emitting diode therapy
  Other Names: Other Names:; LED; Light-emitting diode therapy; LED therapy
  Arms: Placebo light-emitting diode therapy

SUMMARY:
Light-emitting diode Therapy (LEDT) has been used to improve human muscle performance in experimental models and human researches. Now, the investigators used LEDT to increase muscle performance of professional athletes with high performance.

DETAILED DESCRIPTION:
The study assessed muscle performance by vertical jump (height of jump and muscle power); creatine kinase; lactate; metabolism by resonance nuclear magnetic in urine; oxygen uptake (VO2) and its onset kinetic response.

ELIGIBILITY:
Inclusion Criteria:

* professional athletes aged between 14 and 16 years;
* professional athletes aged between 18 and 28 years

Exclusion Criteria:

* previous injury to the femoral quadriceps or hamstring muscles,
* osseous or articular disorder in the lower limbs,
* cardiovascular system disorders,
* systemic disease.

Ages: 14 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Functional performance | 6 weeks
  Muscle performance in vertical jump and running

SECONDARY OUTCOMES:
Biochemical analysis | 1 week
  Blood lactate and creatine kinase assessments

OTHER OUTCOMES:
Aerobic performance | 6 weeks
  oxygen uptake (VO2) and its onset kinetic response.

CONTACTS AND LOCATIONS:
Overall Officials: Cleber Ferraresi, MSc, Principal Investigator — Universidade Federal de Sao Carlos; Nivaldo A Parizotto, PhD, Study Director — Universidade Federal de Sao Carlos; Vanderlei S Bagnato, PhD, Study Director — University of Sao Paulo
Locations (1):
- Federal University of São Carlos, São Carlos, São Paulo, Brazil

REFERENCES:
- [Background] Ferraresi C, de Brito Oliveira T, de Oliveira Zafalon L, de Menezes Reiff RB, Baldissera V, de Andrade Perez SE, Matheucci Junior E, Parizotto NA. Effects of low level laser therapy (808 nm) on physical strength training in humans. Lasers Med Sci. 2011 May;26(3):349-58. doi: 10.1007/s10103-010-0855-0. Epub 2010 Nov 18. PMID 21086010
- [Background] Vieira WH, Ferraresi C, Perez SE, Baldissera V, Parizotto NA. Effects of low-level laser therapy (808 nm) on isokinetic muscle performance of young women submitted to endurance training: a randomized controlled clinical trial. Lasers Med Sci. 2012 Mar;27(2):497-504. doi: 10.1007/s10103-011-0984-0. Epub 2011 Aug 26. PMID 21870127
- [Derived] Ferraresi C, Beltrame T, Fabrizzi F, do Nascimento ES, Karsten M, Francisco Cde O, Borghi-Silva A, Catai AM, Cardoso DR, Ferreira AG, Hamblin MR, Bagnato VS, Parizotto NA. Muscular pre-conditioning using light-emitting diode therapy (LEDT) for high-intensity exercise: a randomized double-blind placebo-controlled trial with a single elite runner. Physiother Theory Pract. 2015 Jul;31(5):354-61. doi: 10.3109/09593985.2014.1003118. Epub 2015 Jan 14. PMID 25585514